CLINICAL TRIAL: NCT00827775
Title: Blood Pressure, Endothelial Cell Dysfunction, and Outcomes in Dialysis Patients
Brief Title: Mechanisms and Treatment of Intradialytic Hypertension
Acronym: MATCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Peter Van Buren, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102008-042; NIH K23 HL092297
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Intradialytic Hypertension
Keywords: Hypertension; Hemodialysis
MeSH Terms: conditions — Hypertension | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients without intradialytic hypertension defined as average pre to post hemodialysis SBP falling >10 mmhg for more than 4/6 of the last dialysis treatment sessions
- Intervention (Active Comparator): Patients with intradialytic hypertension defined as average pre to post hemodialysis SBP elevation of >10 mmhg for more than 4/6 of the last dialysis treatment sessions
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol 6.25 mg BID titrated weekly to maximum of 50 mg bid
  Arms: Intervention

SUMMARY:
1. To determine in a cross sectional case-controlled cohort study of 50 hemodialysis patients if blood pressure elevations with hemodialysis are associated with decreased endothelial cell function (measured by brachial artery flow mediated dilation and endothelial progenitor cell number), both of which are novel mechanistic markers in the causal pathway for detrimental cardiovascular outcomes; and
2. To determine if lowering blood pressure with carvedilol in 25 ESRD subjects with blood pressure elevations with hemodialysis can improve endothelial cell dysfunction as a surrogate mechanistic marker for improving cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* on hemodialysis > 30 days
* aged 18 to 80 years old
* ability to provide informed consent
* Primary nephrologist deems patient is at target dry weight
* Predialysis SBP >140 or postdialysis SBP>130

Exclusion Criteria:

* Patients with active wounds
* Blood pressure unable to be measured by routine mechanisms in the upper extremity
* Change in blood pressure medications in the previous 2 weeks
* Intolerance of beta or alpha-blockers
* pregnancy
* Resting heart rate <50
* Life expectancy < 6 months
* Current therapy with carvedilol or contraindication to carvedilol (ONLY in the intervention arm)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jula K Inrig, MD, MHS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - UTSW Oakcliff Davita Dialysis, Dallas, Texas
  - UTSW Dallas East Davita Dialysis (Buckner unit), Dallas, Texas
  - UTS Dallas Dialysis (Elmbrook), Dallas, Texas

REFERENCES:
- [Result] Inrig JK, Van Buren P, Kim C, Vongpatanasin W, Povsic TJ, Toto R. Probing the mechanisms of intradialytic hypertension: a pilot study targeting endothelial cell dysfunction. Clin J Am Soc Nephrol. 2012 Aug;7(8):1300-9. doi: 10.2215/CJN.10010911. Epub 2012 Jun 14. PMID 22700888
- [Result] Inrig JK, Van Buren P, Kim C, Vongpatanasin W, Povsic TJ, Toto RD. Intradialytic hypertension and its association with endothelial cell dysfunction. Clin J Am Soc Nephrol. 2011 Aug;6(8):2016-24. doi: 10.2215/CJN.11351210. Epub 2011 Jul 14. PMID 21757643
- [Result] Van Buren PN, Kim C, Toto R, Inrig JK. Intradialytic hypertension and the association with interdialytic ambulatory blood pressure. Clin J Am Soc Nephrol. 2011 Jul;6(7):1684-91. doi: 10.2215/CJN.11041210. PMID 21734087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 25 | 30
Completed | 25 | 25
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (7.9) | 53.9 (11.1) | 54.5 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 31
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Progenitor Cells
Description: 1. ALDH bright cells reported as percentage of mononuclear cells. These were assayed using flow cytometry
  2. CD34/CD133 endothelial progenitor cells reported as percentage of mononuclear cells. These were assayed using flow cytometry
Time Frame: 12 weeks
Population: Follow up measurements were only obtained in the intervention subjects receiving carvedilol
Measure: Median (Inter-Quartile Range); unit: % of mononuclear cells
Arm/Group | Control | Intervention
Number analyzed (Participants) | 25 | 25
% of mononuclear cells
  Baseline ALDH bright | 0.052 [0.042 to 0.076] | 0.034 [0.017 to 0.08]
  Follow up ALDH bright: number analyzed (Participants) | 0 | 25
  Follow up ALDH bright |  | 0.027 [0.013 to 0.048]
  Baseline CD34/CD133 endothelial progenitor cells | 0.059 [0.036 to 0.070] | 0.033 [0.016 to 0.051]
  Follow up CD34/CD133: number analyzed (Participants) | 0 | 25
  Follow up CD34/CD133 |  | 0.029 [0.019 to 0.049]

2. Secondary Outcome: Flow Mediated Vasodilation
Description: Measured as percent change in brachial artery diameter from baseline to post shear stress for an individual measurement. Follow up measurements were obtained in intervention subjects 12 weeks later
Time Frame: 12 weeks
Population: Follow up measurements were only obtained in intervention subjects receiving carvedilol
Measure: Mean (Standard Deviation); unit: % dilation from baseline
Arm/Group | Control | Intervention
Number analyzed (Participants) | 25 | 25
% dilation from baseline
  Baseline FMD | 1.67 (1.24) | 1.03 (0.7)
  Follow Up FMD: number analyzed (Participants) | 0 | 25
  Follow Up FMD |  | 1.4 (0.84)

ADVERSE EVENTS:
Time Frame: First day of enrollment to end of study, an average 12 weeks
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 5/25
Other Adverse Events (participants affected / at risk) | 0/25 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=25) | Intervention (N=25)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemodialysis Access Revision (Vascular disorders) | 0 (0) | 1 (1)
Fluid Overload (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=25) | Intervention (N=25)
Symptomatic Intradialytic Hypotension (Cardiac disorders) | 0 (0) | 22 (22) — There were 22 episodes total out of 920 dialysis treatments among the 25 patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No